CLINICAL TRIAL: NCT03595332
Title: Addressing Health Disparities in Childhood Obesity, One Summer at a Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Arizona University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 1193689; U54MD012388 (NIH)
Record Dates: First submitted 2018-06-22; First posted 2018-07-23 (Actual); Results first posted 2022-09-29 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention (Experimental): Summer activity program: Children will receive the summer scorecard program during the first summer of the 2-year study.
  Interventions: Other: Summer activity program
- Delayed intervention (Experimental): Summer activity program: Children will receive the summer scorecard program during the second summer of the 2-year study.
  Interventions: Other: Summer activity program

INTERVENTIONS:
Other: Summer activity program — Children receive a summer scorecard to facilitate access to local facilities for exercise.

SUMMARY:
Almost 50% of Native American and Hispanic children are overweight or obese by the 5th grade. Research has demonstrated that the 'obesity gap' facing minority students is largely due to summer weight gain. However, very few summer programs have been tested among these populations. To encourage summer physical activity, the CDC developed a program that partners with local businesses to provide children with a 'scorecard' of subsidized or free local activities. The program has not been tested among Hispanic or Native American children. This study aims to test the impact of the scorecard program on Body Mass Index percentile, physical activity, sedentary behavior, barriers to physical activity and self-efficacy.

DETAILED DESCRIPTION:
Over 50% of Native American children are overweight or obese by 5th grade, with similar rates found among Hispanics. Native American children have been estimated to have 9 times the diabetes rates of non-Hispanic Whites, suggesting an impending public health crisis without action. Recent research has demonstrated that the 'obesity gap' facing minority students is largely due to summer weight gain, with rapid increases ages 7-11. However, statewide in Arizona, only 22% of children participate in summer activities, despite 65% of parents expressing interest. Thus, we know which populations are at highest risk, at what developmental age changes occur most rapidly and that interventions are most needed in the summer, but that this need is not being met. A modest amount of research has evaluated summer programming, but almost none among Native Americans/Hispanics.

In 2004, the CDC developed a 'Summer Scorecard' intervention, a partnership with local businesses to provide children with a 'scorecard' of subsidized or free local activities. The Summer Scorecard program has not been tested among Hispanic and Native American children. Therefore, the current study propose to assess the effectiveness of the VSS among children ages 7-11 in the 4 highest risk elementary schools in the study area utilizing a randomized design. Two schools will participate in the first summer, and the remaining two children will participate in the second summer. Primary outcomes include objectively measured participation, body composition (BMI percentile), physical activity, sedentary behavior, reported barriers to physical activity and self-efficacy using survey instruments previously developed and tested by the Centers for Disease Control and Prevention. It is hypothesized that children participating in the summer program will increase their physical activity, self-efficacy, reduce their reported barriers to physical activity. In addition, it is hypothesized that they will show reduction in BMI percentile score compared to averages in their school and the school district.

ELIGIBILITY:
Inclusion Criteria:

* Children who are enrolled in one of the 4 high-risk schools in 2nd through 5th grade, whose parents/legal guardians provide consent and provide assent.

Exclusion Criteria:

* Children who are not enrolled in the selected schools, or whose parents/legal guardians do not provide consent, or whom do not provide assent.

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fit kids of Arizona, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huhman ME, Potter LD, Duke JC, Judkins DR, Heitzler CD, Wong FL. Evaluation of a national physical activity intervention for children: VERB campaign, 2002-2004. Am J Prev Med. 2007 Jan;32(1):38-43. doi: 10.1016/j.amepre.2006.08.030. PMID 17218189
- [Background] Huhman M, Potter LD, Wong FL, Banspach SW, Duke JC, Heitzler CD. Effects of a mass media campaign to increase physical activity among children: year-1 results of the VERB campaign. Pediatrics. 2005 Aug;116(2):e277-84. doi: 10.1542/peds.2005-0043. PMID 16061581

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Intervention | Delayed Intervention
Started | 92 | 130
Completed | 76 | 106
Not Completed | 16 | 24
Not completed — Lost to Follow-up | 16 | 22
Not completed — Unable to retrieve ID from school | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Intervention | Delayed Intervention | Total
Number analyzed (Participants) | 92 | 130 | 222
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 92 | 130 | 222
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.80 (1.86) | 9.29 (1.61) | 9.09 (1.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 57 | 113
  Male | 36 | 73 | 109
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 15 | 40 | 55
  Race/Ethnicity: Hispanic | 42 | 42 | 84
  Race/Ethnicity: American Indian/Alaskan Native | 25 | 47 | 72
  Race/Ethnicity: Native Hawaiian/Pacific Islander | 1 | 0 | 1
  Race/Ethnicity: Black | 0 | 1 | 1
  Race/Ethnicity: Two or more | 5 | 0 | 5
  Race/Ethnicity: Unknown | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 92 | 130 | 222
Baseline BMI% [Mean (Standard Deviation); unit: Percentile] | 59.53 (30.08) | 66.23 (32.02) | 63.43 (31.32)

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index Percentile Score Change at 10 Weeks
Description: Body mass index (BMI) will be calculated as kg/m2 and BMI-percentile score calculated using the L, M, S parameters published by the Centre for Disease Control and Prevention. BMI Percentile-score are measures of relative weight adjusted for child age and sex. The percentile indicates value relative to reference populations for age and sex, with at or below 5th percentile indicating the child being underweight, between 5 and 85th percentile as having a healthy weight, 85th to 95th percentile as being overweight and 95th percentile and above indicative of having obesity.
Time Frame: Measured at baseline and 10-weeks after baseline
Measure: Mean (Standard Deviation); unit: Percentile
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 76 | 106
Percentile | 0.307 (0.967) | 1.755 (1.560)
Statistical Analysis 1: Comparison: Immediate Intervention vs Delayed Intervention; Test type: Equivalence — The analysis tests whether for both groups combined, the baseline to 10-week follow-up BMI percentile scores are significantly different from zero; p = 0.248, Regression, Linear — This test compares baseline to 10-week post-test for both groups combined, to test the null hypothesis that the BMI Percentile score would not be different from zero. A p-value of 0.05 was used as a priori threshold for statistical significance; Linear regression with Generalized Estimating Equations to account for nested data structure of 222 children nested within 150 families and 4 schools; Mean Difference (Final Values) = 1.137, 95% CI 2-sided [-0.793 to 3.067], Standard Error of Mean 0.9846

2. Primary Outcome: Overweight Participants Body Mass Index Percentile Score Change
Description: Body mass index (BMI) will be calculated as kg/m2 and BMI percentile calculated using the L, M, S parameters published by the Centre for Disease Control and Prevention. BMI percentiles are measures of relative weight adjusted for child age and sex. This analysis includes only those children who were overweight by CDC standards (equal or greater to 85th percentile for age and sex), as they were the high-risk group of interest for the study.
Time Frame: Baseline to 10 weeks
Population: This analysis includes only those children who were overweight by CDC standards (equal or greater to 85th percentile for age and sex), as they were the high-risk group of interest for the study.
Measure: Mean (Standard Error); unit: Percentile
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 23 | 54
Percentile | -2.632 (1.594) | -3.444 (1.836)
Statistical Analysis 1: Comparison: Immediate Intervention vs Delayed Intervention; Test type: Equivalence — Analysis tested whether BMI Percentile score change among overweight participants (BMI equal or greater than 85th percentile at baseline) significantly changed from baseline to follow-up (was significantly different from zero). This was a subset analysis among the highest risk participants in the study; p = 0.018, Regression, Linear — The p-value threshold was 0.05 for all comparisons; Linear regression with Generalized Estimating Equations to account for nested data structure of children within schools and families; Mean Difference (Final Values) = -3.173, 95% CI 2-sided [-5.806 to -0.541], Standard Error of Mean 1.34 — A negative parameter suggests a decreased BMI Percentile

3. Secondary Outcome: Body Mass Index Percentile Score Change at 1 Year
Description: Body mass index (BMI) will be calculated as kg/m2 and BMI-Percentile score calculated using the L, M, S parameters published by the Centre for Disease Control and Prevention. BMI Percentile-score are measures of relative weight adjusted for child age and sex.
Time Frame: Measured 1-year after baseline
Population: The delayed intervention group 1-year BMI Percentile follow-up was not possible as all schools closed in March 2020 with no measurements allowed over the next year. Of the 76 children (of 92 total) in the immediate intervention group who completed any follow-up measurements, 64 completed 1-year measurements.
Measure: Mean (Standard Error); unit: Percentile
Groups:
- Delayed Intervention: Summer activity program received during Summer 2.
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 64 | 0
Percentile | 0.363 (1.676) |
Statistical Analysis 1: Comparison: Immediate Intervention vs Delayed Intervention; Test type: Equivalence — Analysis tested the difference in BMI percentile between baseline and 1-year follow-up among participants in the immediate intervention group to test the null hypothesis that no change occurred; p = 0.829, Regression, Linear — A prior threshold for statistical significance was 0.05. No adjustment for multiple comparisons was made; Analysis included Generalized Estimating Equations with linear response variable, accounting for nested data structure; Mean Difference (Final Values) = 0.363, 95% CI 2-sided [-2.922 to 3.648], Standard Error of Mean 1.676

4. Secondary Outcome: Change in Intention to Engage in Physical Activity From Baseline to 10 Weeks
Description: During your free time on most days, how likely will you do physical activities? with Likert type 5-answer options (1,2,3,4 or 5) ranging from (1) "I will not be active" to (5) "For sure I will be active". The minimum score is 1, maximum score is 5. Higher scores mean greater intentions to engage in physical activity.
Time Frame: Measured at baseline and at 10-weeks (after summer program)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 76 | 106
score on a scale | 0.238 (0.222) | 0.311 (0.154)
Statistical Analysis 1: Comparison: Immediate Intervention vs Delayed Intervention; Test type: Equivalence — Analysis test whether for both groups combined, Baseline to 10-week change in reported intention of physical activity was significantly different from zero; p = 0.026, Regression, Linear — A priori threshold for statistical significance is 0.05. No adjustments for multiple comparisons were made; Linear regression models with Generalized Estimating Equations to account for nested data were made; Mean Difference (Final Values) = 0.284, 95% CI 2-sided [0.034 to 0.534], Standard Error of Mean 0.128 — A positive parameter would suggest an increase in intentions to be physically active

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Immediate Intervention: Immediate Group: Summer activity program: Children received the summer scorecard program during the first summer of the 2-year study.
  Summer activity program: Children received a summer scorecard to facilitate access to local facilities for exercise.
- Immediate Intervention: Delayed Group: The Delayed intervention group did not receive any intervention during the first summer of the 2-year study.
- Delayed Intervention: Immediate Group: The Immediate intervention group did not receive any intervention during the second summer of the 2-year study.
- Delayed Intervention: Delayed Group: Summer activity program: Children received the summer scorecard program during the second summer of the 2-year study.
  Summer activity program: Children received a summer scorecard to facilitate access to local facilities for exercise.
Arm/Group | Immediate Intervention: Immediate Group | Immediate Intervention: Delayed Group | Delayed Intervention: Immediate Group | Delayed Intervention: Delayed Group
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/130 | 0/92 | 0/130
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/130 | 0/92 | 0/130
Other Adverse Events (participants affected / at risk) | 0/92 | 0/130 | 0/92 | 0/130

LIMITATIONS AND CAVEATS:
Limitations include a specific setting in the Southwestern United States. Second, any dose-response analyses were reliant on self-report. Loss to follow-up, likely due to children moving schools, reduced the final sample from 222 to 186 with at least partial follow-up measures (178 completed). Finally, COVID-19 prevented collection of secondary outcome 1-year follow-up BMI Percentile (Apr 2020) for one group as the school district shut down (and remote for a year after reopening).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-04-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT03595332/Prot_002.pdf
  • Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT03595332/SAP_003.pdf
  • Informed Consent Form (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT03595332/ICF_001.pdf